CLINICAL TRIAL: NCT00075855
Title: The Use of Low Dose Testosterone To Enhance Libido In Female Cancer Survivors: A Phase III Randomized, Placebo-Controlled, Double-Blind Crossover Study
Brief Title: Low-Dose Testosterone in Improving Libido in Postmenopausal Female Cancer Survivors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N02C3; NCI-2012-02568 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000349426 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-01-09; First posted 2004-01-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Cancer Survivor; Sexual Dysfunction; Sexuality and Reproductive Issues; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: sexual dysfunction; unspecified adult solid tumor, protocol specific; sexuality and reproductive issues; cancer survivor
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Sexuality | interventions — Testosterone Propionate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- testosterone (Experimental): Patients receive topical testosterone once daily for 4 weeks. After 4 weeks, patients cross over to the other treatment arm.
  Changes in sexual functioning, mood states, and medical outcome vitality are assessed at baseline and then at the end of weeks 4 and 8.
  Patients who continue or restart testosterone cream after the 8-week study period are followed at 6 months.
  Interventions: Drug: therapeutic testosterone
- placebo (Other): Patients receive a topical placebo once daily for 4 weeks. After 4 weeks, patients cross over to the other treatment arm.
  Changes in sexual functioning, mood states, and medical outcome vitality are assessed at baseline and then at the end of weeks 4 and 8.
  Patients who continue or restart testosterone cream after the 8-week study period are followed at 6 months.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: therapeutic testosterone
  Arms: testosterone
Other: placebo
  Arms: placebo

SUMMARY:
RATIONALE: The hormone testosterone may improve the libido (sex drive) in women. It is not yet known whether testosterone is effective in improving libido in female cancer survivors.

PURPOSE: This randomized phase III trial is studying how well low-dose testosterone works to improve libido in postmenopausal cancer survivors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of low-dose testosterone, in terms of average intra-patient change in libido, in postmenopausal female cancer survivors with a decreased libido.

Secondary

* Determine the toxic effects of this drug in these patients.
* Determine the levels of estrogen and testosterone and SGOT in patients reporting a decreased libido before and after treatment with this drug.
* Determine whether increasing libido significantly positively affects pleasure from sexual activity in patients treated with this drug.
* Determine the effect of this drug on vitality, general quality of life, and overall mood in these patients.

OUTLINE: This is a double-blind, placebo-controlled, randomized, crossover, multicenter study. Patients are stratified according to antidepressant medication use (yes vs no), age (under 50 vs 50 to 60 vs 61 to 70 vs over 70), tamoxifen or other selective estrogen receptor modulator use (yes vs no), and ovarian status (in place [natural menopause or hysterectomy] vs not in place [bilateral oophorectomy]). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive topical testosterone once daily for 4 weeks.
* Arm II: Patients receive a topical placebo once daily for 4 weeks. After 4 weeks, patients cross over to the other treatment arm.

Changes in sexual functioning, mood states, and medical outcome vitality are assessed at baseline and then at the end of weeks 4 and 8.

Patients who continue or restart testosterone cream after the 8-week study period are followed at 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* History of cancer

  * No active disease
* Currently has a sexual partner
* Reports a decrease in sexual desire or libido and would like an intervention for it

  * Defined as a score of less than 8 on the numerical analogue scale

PATIENT CHARACTERISTICS:

Age

* See Menopausal status

Sex

* Female

Menopausal status

* Postmenopausal, defined as the following:

  * Surgically induced menopause OR absence of a period for at least 12 months (naturally or treatment-induced)

Performance status

* ECOG 0-1

Hematopoietic

* WBC ≥ 2,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL
* No untreated anemia

Hepatic

* SGOT ≤ 1.5 times upper limit of normal (ULN)
* No known liver disease

Renal

* Creatinine ≤ 1.5 times ULN
* No renal dysfunction

Cardiovascular

* No coronary artery disease
* No congestive heart failure

Other

* No untreated hypothyroidism
* No diabetes
* No major depressive disorder requiring treatment

PRIOR CONCURRENT THERAPY:

Chemotherapy

* Concurrent cytotoxic chemotherapy (e.g., tamoxifen or aromatase inhibitors) allowed

Endocrine therapy

* No prior testosterone
* No prior androgen agents for libido
* Concurrent selective estrogen receptor modulators allowed
* Concurrent vaginal estrogen allowed provided it was initiated ≥ 1 month ago and continued at the same dose during study participation

Radiotherapy

* Concurrent radiotherapy allowed

Surgery

* No prior major pelvic surgery resulting in anatomical changes to the vaginal anatomy

  * Prior hysterectomy allowed

Other

* Concurrent antidepressants for postmenopausal mood or hot flashes allowed provided patient is on a stable dose that will not change within the next 8 weeks
* No concurrent anticoagulants or propanolol

  * Concurrent anticoagulants for central or peripheral line maintenance (e.g., warfarin 1 mg daily or heparin flushes) allowed
* No other concurrent treatment for decreased libido

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2004-04; Primary Completion 2007-05 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Overall mood | Up to 6 months

SECONDARY OUTCOMES:
quality of life | Up to 6 months
overall vitality | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Loprinzi, MD — Mayo Clinic
Locations (16):
- United States (16):
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - CCOP - Dayton, Dayton, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin

REFERENCES:
- [Background] Jones B, Haughie S. Re: randomized controlled trial to evaluate transdermal testosterone in female cancer survivors with decreased libido: north central cancer treatment group protocol N02C3. J Natl Cancer Inst. 2008 Oct 15;100(20):1482; author reply 1482. doi: 10.1093/jnci/djn311. Epub 2008 Oct 7. No abstract available. PMID 18840823
- [Result] Barton DL, Wender DB, Sloan JA, Dalton RJ, Balcueva EP, Atherton PJ, Bernath AM Jr, DeKrey WL, Larson T, Bearden JD 3rd, Carpenter PC, Loprinzi CL. Randomized controlled trial to evaluate transdermal testosterone in female cancer survivors with decreased libido; North Central Cancer Treatment Group protocol N02C3. J Natl Cancer Inst. 2007 May 2;99(9):672-9. doi: 10.1093/jnci/djk149. PMID 17470735